CLINICAL TRIAL: NCT07387848
Title: A Phase II,Open Label, Single Arm, Multicenter Study Investigating the Efficacy and Safety of Glofitamab When Used as a Bridge to and/or Consolidation Post-transplant for Patients With Relapsed/Refractory B-cell Lymphomas Transformed Low Grade B Cell Lymphoma) Fit and Eligible for ASCT
Brief Title: Glofitamab as a Bridge to and/or Consolidation Post Autologous Stem Cell Transplant in Patients With Relapsed B Cell Lymphomas
Acronym: GLO-PACT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIO-2025-0317
Record Dates: First submitted 2026-01-19; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Diffuse Large B Cell Lymphoma Refractory
Keywords: Glofitamab; DLBCL; Relapse; Refractory; ASCT
MeSH Terms: conditions — Recurrence | interventions — glofitamab

STUDY DESIGN:
Intervention Model Description: This is an investigator initiated open label, single arm, multicenter, phase II trial investigating the efficacy and safety of Glofitamab when used as a bridge to and/or consolidation post-transplant for patients with relapsed/refractory B-cell lymphomas (DLBCL or transformed low grade B cell lymphoma) fit and eligible for ASCT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- single arm study assessing the efficacy and safety of Glofitamab as a bridge to and/or consolidation (Experimental): Participants who complete two cycles of Rituximab-chemotherapy will undergo evaluation by PET scan.
  * Complete responders will proceed to a third cycle of Rituximab-chemotherapy, followed by autologous stem cell transplantation (ASCT) and six cycles of consolidation Glofitamab.
  * Participants with an incomplete response will receive three cycles of salvage Glofitamab, after which they will be re-evaluated by PET scan. Patients achieving a complete response at this stage will proceed to ASCT, followed by three cycles of consolidation Glofitamab. Non-responders will be discontinued from the study
  Interventions: Drug: Glofitamab

INTERVENTIONS:
Drug: Glofitamab — Glofitamab is started with initially a step-up dosing of 2.5 mg on C1D1 then 10 mg on C1D8 to be followed by 30 mg every 3 weeks for a total of 3 cycles. Disease evaluation is repeated after completion of 3 cycles of Glofitamab, and patients achieving PR or better then undergo ASCT followed by 3 cycles post consolidation glofitamab (30 mg every 3 weeks).

SUMMARY:
This is an investigator-initiated, open-label, single-arm, multicenter, Phase II clinical study. The study is designed to evaluate the safety and potential effectiveness of glofitamab in adults with their disease, diffuse large B-cell lymphoma (DLBCL has either not responded to initial treatment or has returned after an initial response and who are eligible and medically fit for autologous stem cell transplantation (ASCT). Autologous stem cell transplantation is a commonly used treatment in this situation and involves high-dose chemotherapy followed by infusion of your own stem cells, which are collected from your blood several weeks before the transplant.

The purpose of this study is to assess glofitamab, which is not part of standard treatment. Glofitamab is a type of antibody designed to attach to both lymphoma cells and certain immune cells called T cells. By bringing these cells together, glofitamab may help activate the immune system so that T cells can better recognize and destroy lymphoma cells. In this study, glofitamab may be used as a "bridge" to transplantation and/or as consolidation treatment after the transplant, depending on how the disease responds to chemotherapy given before the transplant.

In recent years, newer immune-based treatments such as CAR-T cell therapy have shown benefit for patients whose lymphoma does not respond to or returns after chemotherapy. CAR-T therapy involves collecting immune cells, modifying them in a laboratory, and then reinfusing them into the patient. However, access to CAR-T therapy is limited in some regions, including Lebanon, and autologous stem cell transplantation remains an important treatment option

DETAILED DESCRIPTION:
This is an investigator initiated open label, single arm, multicenter, phase II trial investigating the efficacy and safety of Glofitamab when used as a bridge to and/or consolidation post-transplant for patients with relapsed/refractory B-cell lymphomas (DLBCL or transformed low grade B cell lymphoma) fit and eligible for ASCT.

Primary Objective: To evaluate the efficacy of glofitamab when used as a bridge to and/or consolidation post-transplant for patients with relapsed/refractory B-cell lymphomas (DLBCL or transformed low grade B cell lymphoma) fit and eligible for ASCT ,

Secondary Objectives:

* To evaluate the efficacy of glofitamab when used as a bridge to and/or consolidation post-ASCT.
* To evaluate the safety and tolerability of glofitamab in this setting
* To evaluate the effect of glofitamab when used as a bridge to and/or consolidation post ASCT on health-related quality of life (HRQoL) Exploratory Objectives
* To evaluate the effect of treatment with glofitamab on acute phase reactants such as fibrinogen and its clinical significance.

Adult patients (age 18-65) with primary refractory disease or relapsed CD20-positive DLBCL (all subtypes including primary mediastinal B cell lymphoma, high grade B cell lymphoma, large B cell lymphoma etc) or transformed low grade B-cell lymphoma, who are eligible for ASCT, planned to receive salvage therapy with Rituximab-chemotherapy regimens followed by ASCT.

ELIGIBILITY:
Inclusion Criteria:

- To be eligible to participate in this trial, an individual must meet all of the following criteria:

1. Provision of signed and dated informed consent form (ICF) ) by the patient/impartial witness/legal representative before any trial related procedures.
2. Male or female aged between 18 and 65 years.
3. Ability and willingness to comply with the study protocol.
4. Histologically confirmed diagnosis of primary refractory or relapsed DLBCL (all subtypes including primary mediastinal B cell lymphoma, high grade B cell lymphoma, large B cell lymphoma etc) or transformed low grade B cell lymphoma planned for salvage Rituximab-chemotherapy regimens followed by ASCT.
5. Patients with a life expectancy of at least 6 months.
6. All patients must be stable without any signs of active infection, systemic (oral or parenteral) corticosteroid or anticonvulsant therapy for at least 2 weeks prior to study treatment. Inhaled non-absorbable and topical corticosteroid use are permitted as indicated.
7. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1 with no deterioration over the previous 2 weeks.
8. Women of child-bearing potential and male subjects shall agree to take medically acceptable contraception measures while on study treatment and for 3 months following completion of study treatment. All women of child-bearing potential must have a negative blood pregnancy test at screening.

   Women must remain abstinent or use contraceptive methods with a failure rate of ≤1% per year during the study treatment period and for 2 months after the final dose of glofitamab, 3 months after the final dose of tocilizumab (if applicable), 12 months after rituximab or chemotherapy, or 18 months after the final dose of obinutuzumab. Women must refrain from donating eggs during this same period. A woman is considered of childbearing potential if she is postmenarchal, has not reached a postmenopausal state (≥12 continuous months of amenorrhea with no identified cause other than menopause), and is not permanently infertile due to surgery (i.e., removal of ovaries, fallopian tubes, and/or uterus) or another cause as determined by the investigator (i.e., Müllerian agenesis). The definition of childbearing potential may be adapted for alignment with local guidelines or regulations. Examples of contraceptive methods with a failure rate of ≤1% per year include bilateral tubal ligation, male sterilization, hormone-releasing intrauterine devices, and copper intrauterine devices. Hormonal contraceptive methods must be supplemented by a barrier method. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the individual. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post ovulation methods) and withdrawal are not adequate methods of contraception. If required per local guidelines or regulations, locally recognized adequate methods of contraception and information about the reliability of abstinence will be described in the local Informed Consent Form. For men who are not surgically sterile (or with azoospermia for other reasons): Investigators will discuss sperm conservation prior to initiation of study treatment for male participants. Participants who agree to remain abstinent (refrain from heterosexual intercourse) or use contraception, and agree to refrain from donating sperm, as defined below: With a female partner of childbearing potential who is not pregnant, men must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of ≤1% per year during the study treatment period and for 2 months after the final dose of glofitamab, 3 months after the final dose of tocilizumab (if applicable), 6 months after rituximab, ICE (ifosfamide, carboplatin, and etoposide) or obinutuzumab. Men must refrain from donating sperm during this same period. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the individual. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post ovulation methods) and withdrawal are not adequate methods of contraception. If required per local guidelines or regulations, locally recognized adequate methods of contraception and information about the reliability of abstinence will be described in the local Informed Consent Form.
9. Patients with at least one bi-dimensionally measurable (≥1.5 cm) nodal lesion, or one bi-dimensionally measurable (≥1 cm) extranodal lesion, as measured on CT scan.
10. Adequate hematologic function (unless attributable to the underlying disease, as established by extensive bone marrow involvement or associated with hypersplenism secondary to the involvement of the spleen by DLBCL per the investigator), defined as follows:

    - ANC ≥1.0 x109/L ( ≥1000/μL) Participants with a history of benign ethnic neutropenia may be included with ANC ≥0.75x109/L (≥750/μL).

    - Platelet count ≥50x109/L (≥50,000/μL) without a transfusion in the week prior to starting study treatment.
11. Adequate renal function, defined as an estimated CrCl ≥ 45 mL/min.
12. Participants who have a negative HIV test at screening, with the following exception: Individuals with a positive HIV test at screening are eligible provided they are stable on anti-retroviral therapy for at least 4 weeks, have a CD4 count ≥200/μL, have an undetectable viral load, and have not had a history of opportunistic infection attributable to AIDS within the last 12 months.

Exclusion Criteria:

* An individual, who meets ANY of the following criteria, will be excluded from participation in this trial:

  1. Patients receiving any investigational drug, biological, immunological therapy within the previous 21 days before enrollment.
  2. Presence of any severe or uncontrolled systemic disease or condition, including serious cardiac, pulmonary or renal conditions; any type of bacterial, viral, fungal or other infection that would pose a significant risk to the patient in the opinion of the investigator; or active Hepatitis B or positive HCV antibodies.
  3. Any unresolved toxicities from prior therapy, greater than CTCAE-version 5 grade 2 at the time of starting study treatment, with exception of alopecia.
  4. Patients with a significant cardiovascular disease or condition, including any of the following:

     1. Congestive heart failure (CHF) currently requiring therapy and patients with New York Heart Association Class III/IV CHF
     2. LVEF < 50%
     3. Need for antiarrhythmic medical therapy for a ventricular arrhythmia or patients with uncontrolled or unstable cardiac arrhythmias
     4. Severe conduction disturbance (e.g., second- or third-degree AV block)
  5. Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values:

     1. Absolute neutrophil count < 1 x 109/L (or < 0.75 x 109/L in case of ethnic neutropenia due to excess margination)
     2. Platelet count < 50 x 109/L (Transfusion-dependent patients are excluded)
  6. Severe hepatic and/or renal impairment as demonstrated by any of the following:

     a. Alanine aminotransferase > 2.5 times the upper limit of normal (ULN) b. Aspartate aminotransferase > 2.5 times ULN c. Total bilirubin > 1.5 times ULN (Total bilirubin >3 times the ULN in patients with documented Gilbert's Syndrome (unconjugated hyperbilirubinemia) d. Creatinine clearance < 45 mL/min (measured or calculated by Cockcroft and Gault equation). Confirmation of creatinine clearance is only required when creatinine is >1.5 times ULN
  7. Judgement by the investigator that the patient should not participate in the study if the patient is unlikely to comply with all study procedures and treatment.
  8. Significant medical or psychiatric illness that would interfere with compliance and ability to tolerate treatment as outlined in the protocol.
  9. History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies (or recombinant antibody-related fusion proteins) or known sensitivity or allergy to murine products.
  10. The presence of any contraindication to: Obinutuzumab, rituximab, or tocilizumab.
  11. Prior treatment with glofitamab or other bispecific antibodies targeting both CD20 and CD3.

  10. Peripheral neuropathy assessed to be Grade >1 according to National Cancer Institute (NCI) CTCAE) v5.0 at Enrollment.

  11. Current or history of CNS disease, such as stroke, epilepsy, CNS vasculitis, o neurodegenerative disease (note: Participants with a history of stroke who have not experienced a stroke or transient ischemic attack within the past 2 years and have no residual neurologic deficits, as judged by the investigator, are allowed).

  12. Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment or any major episode of infection (as evaluated by the investigator) within 2 weeks prior to the first study treatment. 13. History of other malignancy that could affect compliance with the protocol or interpretation of results, with the following exceptions:

Note:

* Participants with a history of curatively treated basal or squamous cell carcinoma of the skin or in situ carcinoma of the cervix at any time prior to enrollment are allowed.
* Participants with low-grade, early-stage prostate cancer (Gleason score 6 or below, Stage 1 or 2 with no requirement for therapy at any time prior to enrollment are allowed.
* Participants with any other malignancy appropriately treated with curative intent and the malignancy has been in remission without treatment for ≥ 2 years prior to enrollment are eligible.
* Participants receiving adjuvant endocrine therapy for non-metastatic, hormone receptor positive breast cancer for ≥2 years prior to enrollment are eligible.

  14. Contraindications to treatment with rituximab, Obinutuzumab or tocilizumab.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-04-15 (Estimated); Primary Completion 2031-12-15 (Estimated); Study Completion 2031-12-15 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of glofitamab when used as a bridge to and/or consolidation post-transplant for patients with relapsed/refractory B-cell lymphomas (DLBCL or transformed low grade B cell lymphoma) fit and eligible for ASCT | 3 years
  Progression free survival (PFS) at 1 year post relapse-defined as the time from infusion of first salvage chemotherapy to the first occurrence of disease progression or death from any cause, whichever occurs first as determined by the investigator

SECONDARY OUTCOMES:
To evaluate the 3 years overall survival | 3 years
  Overall survival (OS) at 3 year post relapse defined as the time from first dose of salvage chemotherapy to date of death from any cause
To evaluate the safety and tolerability of glofitamab in this setting | 3 years
  Incidence and severity of adverse events (AEs), with severity determined according to the national Cancer Institute Common Toxicity Criteria for Adverse Events, Version 5.0 (NCI CTCAE v5.0)
To evaluate the effect of glofitamab when used as a bridge to and/or consolidation post ASCT on health-related quality of life (HRQoL) | 3 years
  Changes in QLQ-NHL-HG29 questionnaire results taken before first dose of glofitamab and that taken at end of treatment with glofitamab.
  he EORTC QLQ-NHL-HG29 (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Non-Hodgkin Lymphoma-High-Grade 29) is a disease-specific quality-of-life instrument. Scores are transformed to a 0-100 scale. For functional domains, higher scores indicate better outcomes, whereas for symptom domains, higher scores indicate worse outcomes.
To evaluate the effect of treatment with glofitamab on acute phase reactants such as fibrinogen and its clinical significance | 1 year
  Changes in fibrinogen level from baseline (before starting first dose of glofitamab compared to post each dose of glofitamab and post last dose of glofitamab) will be correlated with PFS and CRS.
To Assess the complete response rate | 1 year
  the complete response (CR) defined as the proportion of patients whose best overall response is CR on positron emission tomography (PET/CT scan) at two time points (at transplant for those receiving glofitamab as a bridge to ASCT, and at end of treatment (EOT) with glofitamab (3-4 weeks after last dose of post-ASCT consolidation with glofitamab) for all patients
To Assess the rate of ASCT | 1 year
  the rate of ASCT is assessed after induction chemotherapy and after 3 doses of Glofitamab for non- responders.
  Rate of ASCT for those receiving Glofitamab as salvage therapy is assessed post induction chemo and post 3 dose Glofitamab for non resposnders.
clinical complete response rate | 6 months
  Rate of complete response (CR) defined as the proportion of patients whose best overall response is CR on positron emission tomography (PET/CT scan) at two time points (at transplant for those receiving glofitamab as a bridge to ASCT, and at end of treatment (EOT) with glofitamab (3-4 weeks after last dose of post-ASCT consolidation with glofitamab) for all patients
Rate of ASCT for patients receiving glofitamab as salvage therapy | 6 months
  The rate of autologous stem cells transplantation of patients who received salvage Glofitamab is defined as the proportion of patients who reached the ASCT after completing the salvage Glofitamab treatment after being evaluated by PET scan and Bone Marrow aspirate and biopsy to confirm complete response rate.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Bazarbachi, MD, Principal Investigator — American University of Beirut Medical Center

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD will be made available upon reasonable request to the study sponsor. Requests must include a research proposal with a clearly defined scientific objective. Access will be subject to sponsor approval and may require execution of a data-sharing agreement, in accordance with applicable ethical and regulatory requirements.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: after publication
Access Criteria: De-identified IPD will be made available upon reasonable request to the study sponsor. Requests must include a research proposal with a clearly defined scientific objective. Access will be subject to sponsor approval and may require execution of a data-sharing agreement, in accordance with applicable ethical and regulatory requirements.